CLINICAL TRIAL: NCT06364761
Title: Assesment of Intermediate and Near Vision After Bag in the Lens Cataract Surgery
Brief Title: Assesment of Intermediate Vision After BIL Cataract Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 24103_BIL_EDOF
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Cataract
Keywords: bag in lens; Intermediate vision
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bag in the lens: Patients who underwent bag in the lens cataract surgery at least 3 months before inclusion in the University Hospital Brussels, Belgium.
  Interventions: Procedure: Bag in the lens cataract surgery

INTERVENTIONS:
Procedure: Bag in the lens cataract surgery — Cataract surgery using the Morcher 89A intraocular lens

SUMMARY:
The goal of this observational study is to learn about the intermediate and near vision in patiënts who underwent cataract surgery with a specific technique, called "bag in the lens".

The main question it aims to answer is whether patiens who underwent this type of cataract surgery have better intermediate vision without spectacle correction than patients who underwent the classic lens in the bag cataract surgery.

Participants will:

* Have to read with and without spectacle correction at different distances (4 meters, 66 centimeters, 40 centimeters)
* Have to fill in 2 questionnaires about visual functioning and spectacle independance

Researchers will compare these values to the same values from the standard population who underwent the classic lens in the bag cataract surgery with a monofocal intraocular lens .

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years old
* Must have underwent bilateral bag in the lens cataract surgery in the University hospital Brussels at least 3 months before inclusion
* Must not meet any exclusion criteria

Exclusion Criteria:

* Prior refractive surgery (other than bag in the lens)
* Glaucoma
* Corneal opacities
* Moderate non proliferative diabetic retinopathy or worse
* Optic neuropathy
* History of uveitis
* Amblyopia
* Residual post-operative astigmatism higher than 1.5 Diopters (D)
* Best corrected visual acuity < 1.0
* Patients unable to cooperate or sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent bilateral bag in the lens cataract surgery in the University Hospital Brussels at least 3 months before inclusion
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intermediate vision | During the only hospital visit required in the study, between april and december 2024
  uncorrected and distance corrected intermediate vision at 66cm in LogMAR

SECONDARY OUTCOMES:
Near vision | During the only hospital visit required in the study, between april and december 2024
  uncorrected and distance corrected intermediate vision at 40cm in LogMAR

CONTACTS AND LOCATIONS:
Overall Officials: Jorgos Koulalis, M.D., Principal Investigator — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: Undecided